CLINICAL TRIAL: NCT00698880
Title: Sequential Preoperative Ipsilateral Hepatic Vein Embolization After Portal Vein Embolization to Induce Further Liver Regeneration in Patients With Hepatobiliary Malignancy
Brief Title: Ipsilateral Hepatic Vein Embolization After Portal Vein Embolization
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Shin Hwang, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Preop_PVE_HVE
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Procedure-Related Complication; Degree of Liver Regeneration
Keywords: Portal vein embolization; Hepatic vein embolization; Liver regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HVE (Active Comparator): Hepatic vein embolization after portal vein embolization
  Interventions: Procedure: Right hepatic vein embolization
- PVE (No Intervention): Only portal vein embolization, historical control group

INTERVENTIONS:
Procedure: Right hepatic vein embolization — Embolization of the right hepatic vein
  Other Names: Sequential right hepatic vein embolization
  Arms: HVE

SUMMARY:
Portal vein embolization (PVE) induces shrinkage of the embolized lobe and compensatory enlargement of the non-embolized lobe, but it does not always induce sufficient liver regeneration. There was no effective method to accelerate liver regeneration in addition to PVE yet.

This study intends to assess the effect of ipsilateral hepatic vein embolization (HVE) performed after Portal vein embolization (PVE) on liver regeneration. During a 1-year study period, preoperative HVE would be performed on 10 or more patients who had shown limited liver regeneration after PVE awaiting right hepatectomy. Sequential application of PVE and HVE may be safe and effective in facilitating contralateral liver regeneration by inducing more severe liver damage than PVE alone.

DETAILED DESCRIPTION:
To prospectively assess the effect of ipsilateral HVE after PVE on liver volume change, this study was designed to continue for 12 months, from March 2007 to February 2008.

This study protocol was approved by our institutional review board, under the condition that, for patient safety, more than one occurrence of accidental coil migration into the heart or lung would lead to study discontinuation. The clinical significance of this risk had not been fully assessed, although it might not be seriously harmful. In addition, informed consent and permission for each PVE and HVE were obtained separately from each patient and/or his/her family members.

The indications for right PVE are patients undergoing right hepatectomy or more extensive liver surgery for hepatobiliary malignancy, but having small FLRs, with mean values less than 40% of total liver volume. Patients with large liver masses are excluded because their parenchymal resection rates were much lower than 60%. For patients with perihilar cholangiocarcinoma, placement of multiple biliary drains was preferred to decompress the entire biliary system, and the timing of PVE was set to when serum total bilirubin level became lower than 5 mg/dL.

The right internal jugular vein was punctured with an 18-gauge needle and a 9-F long sheath (Cook; Bloomington, IN) was inserted. The right hepatic vein (RHV) was selected using a 5-F cobra catheter (Cook) and a 0.035-inch guide wire (Terumo; Tokyo, Japan). Insertion of the guide wire toward the dorsal side was checked with a right lateral view to confirm that it was correctly inserted into the RHV. A 9-F sheath was inserted at the proximal portion of the RHV, followed by placement of a Tulip filter (retrievable vena cava filter; Cook) or a Trap-Ease filter (Cordis; Miami, FL) to prevent migration of deployed coils during embolization of the RHV. The cobra catheter was then advanced into the RHV and the main RHV branches were embolized with coils 8 to 12 mm in diameter (nester embolization coils; Cook).

Multidetector dynamic CT scans were routinely performed before PVE to assess gross liver volume change and tumor progression, and CT scans were performed every week after PVE, HVE, and hepatectomy. All CT images were reconstructed as sections 3 mm thick. The CT images were stored in a Picture Archiving and Communication System (PACS; Petavision; Asan Medical Center, Seoul, Korea), enabling image processing and various measurements including volumetry. In patients undergoing combined caudate resection, the volume of the caudate lobe was not included in the FLR volume. TLV and FLR volume before PVE were used as the baseline liver volumes for liver size comparison.

To assess the histological changes in the livers, 1 cm-sized pieces of liver tissue were excised from the ventral margins of the right posterior section, right anterior section, and left lateral section just after laparotomy. These samples were immediately fixed with 4% paraformaldehyde phosphate solution.

Immunohistochemical stainings were performed using antibody against albumin to assess the synthetic function of the hepatocytes, antibody against proliferating cell nuclear antigen (anti-PCNA) to assess cell replication, and antibody against cleaved caspase-3 to assess apoptosis. Apoptosis was also assayed by terminal deoxynucleotidyl transferase-mediated dUTP-digoxigenin nick-end labeling (TUNEL) staining. Western blots using antibodies against the acute phase proteins TNF-α, caspase-3, Bax, and Bcl-2 were performed to assess the status of proinflammatory cytokine responses. PCNA-positive and caspase-3-positive events were counted in five randomly selected high-power fields on microphotographs.

Specimens for histological examination and histomorphometric analysis were stained with hematoxylin and eosin (H-E). For hepatocyte counts, 10 different HPFs in the same slide were randomly selected.

ELIGIBILITY:
Inclusion Criteria:

* Patients showing small future remnant liver < 40% of whole liver volume

Exclusion Criteria:

* Patients showing small future remnant liver > 40% of whole liver volume
* Inoperable tumor extent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Future remnant left liver volume on multidetector dynamic CT scans | 2 weeks after HVE

SECONDARY OUTCOMES:
Immunohistochemical stainings | during operation

CONTACTS AND LOCATIONS:
Overall Officials: Shin Hwang, MD, PhD, Principal Investigator — Department of Surgery, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea